CLINICAL TRIAL: NCT00085540
Title: A Phase I-II Trial of Depsipeptide in Patients With Recurrent High-Grade Gliomas
Brief Title: FR901228 in Treating Patients With Recurrent High-Grade Gliomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02596; NABTC-0303; U01CA062399 (NIH); CDR0000370817 (Registry Identifier: PDQ (Physician Data Query)); NCT00103909 (obsolete NCT alias)
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Results first posted 2016-11-15 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Adult Anaplastic Astrocytoma; Adult Anaplastic Oligodendroglioma; Adult Giant Cell Glioblastoma; Adult Gliosarcoma; Recurrent Adult Brain Tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Depsipeptides; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase 1 Dose Escalation - Romidepsin (Experimental): Patients receive FR901228 (romidepsin) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Dose escalation two dose levels:
  Romidepsin (depsipeptide): 13.3mg/m2 and 17.7mg/m2
  Pharmacokinetics
  Interventions: Drug: depsipeptide
- Phase 2 Dose from Phase 1 - Romidepsin (Experimental): Patients receive FR901228 (romidepsin) as in phase I at dose level 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Romidepsin (depsipeptide): 13.3mg/m2
  Interventions: Drug: depsipeptide

INTERVENTIONS:
Drug: depsipeptide — Given IV
  Other Names: FK228; FR901228; Istodax; romidepsin

SUMMARY:
This phase I/II trial is studying the side effects and best dose of FR901228 and to see how well it works in treating patients with recurrent high-grade gliomas. FR901228 may stop the growth of tumor cells by blocking the enzymes necessary for their growth

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of FR901228 (depsipeptide) in patients with recurrent malignant gliomas who are taking enzyme-inducing antiepileptic drugs (EIAEDs). (Phase I) II. Determine the safety profile of this drug in these patients. (Phase I) III. Determine the pharmacokinetics and pharmacodynamics of this drug in these patients. (Phase I) IV. Determine the clinical efficacy of this drug, as measured by 6-month progression-free survival and objective tumor response, in these patients. (Phase II) V. Determine the safety profile of this drug when administered at the phase I MTD concurrently with or without EIAEDs in these patients. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study followed by a phase II study. Patients are stratified according to study phase (I vs II), concurrent use of enzyme-inducing anti-epileptic drugs (EIAEDs) (yes vs no), histology (recurrent glioblastoma multiforme/gliosarcoma vs recurrent anaplastic glioma), pre-operative candidacy (yes vs no), and measurable/evaluable disease (yes vs no). Patients are assigned to 1 of 2 treatment groups (group A: no EIAEDs or group B: concurrent use of EIAEDs).

Phase I (group B only): Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of FR901228 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of up to 6 patients experience dose-limiting toxicity.

Phase II (groups A and B):

Group A (phase II): Patients receive FR901228 as in phase I at dose level 1. Group B (phase II): Patients receive FR901228 as in phase I at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Phase I and phase II:

  * Histologically confirmed recurrent intracranial malignant glioma, including any of the following:

    * Glioblastoma multiforme
    * Gliosarcoma
    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Anaplastic mixed oligoastrocytoma
    * Malignant astrocytoma not otherwise specified
* Unequivocal evidence of tumor progression by MRI or CT scan while on a steroid dosage that has been stable for at least 5 days
* Patients previously treated with interstitial brachytherapy or stereotactic radiosurgerymust have confirmation of true progressive disease (rather than radiation necrosis) by positron-emission tomography, thallium scan, magnetic resonance spectroscopy, or surgical documentation
* Must have failed prior radiotherapy that was completed at least 6 weeks ago
* No more than 2 prior therapies (initial treatment and treatment for 1 relapse)*

  * Surgical resection for relapsed disease with no anticancer therapy for up to 12 weeks, followed by a second surgical resection, is considered treatment for 1 relapse
* Patients in group B must have been receiving enzyme-inducing antiepileptic drugs (EIAEDs) for at least the past 2 weeks
* Performance status - Karnofsky 60-100%
* More than 8 weeks
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL (transfusions allowed)
* SGOT < 2 times upper limit of normal (ULN)
* Bilirubin < 2 times ULN
* Creatinine < 1.5 mg/dL
* No congestive heart failure (i.e., New York Heart Association class II-IV, ejection fraction < 40% by MUGA scan or < 50% by echocardiogram and/or MRI)
* No myocardial infarction within the past year
* No uncontrolled dysrhythmias
* No poorly controlled angina
* No significant left ventricular hypertrophy by EKG
* No cardiac ischemia (ST depression of 2 mm) by EKG
* No hypertrophic or restrictive cardiomyopathy from prior treatment or other causes
* No uncontrolled hypertension (i.e., blood pressure ≥ 160/95 mm Hg)
* No cardiac arrhythmia requiring antiarrhythmic medication
* No known cardiac abnormalities (e.g., congenital long QT syndrome and QTc interval > 480 milliseconds)
* No history of sustained ventricular tachycardia, ventricular fibrillation, Torsade de Pointes, or cardiac arrest unless controlled with concurrent automatic implantable cardioverter defibrillator
* No known history of coronary artery disease (e.g., Canadian class II-IV angina)
* No other significant cardiac disease
* No other malignancy within the past 3 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No active infection
* No significant uncontrolled medical illness that would preclude study participation
* No disease that would obscure toxicity or dangerously alter drug metabolism
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 2 weeks after study participation

  * Fertile male patients must continue barrier contraception for 3 months after study participation
* At least 1 week since prior interferon or thalidomide
* No concurrent prophylactic filgrastim (G-CSF)
* No concurrent anticancer immunotherapy
* At least 2 weeks since prior vincristine
* At least 6 weeks since prior nitrosoureas
* At least 3 weeks since prior procarbazine
* No prior FR901228 (depsipeptide)
* No other concurrent anticancer chemotherapy
* See Disease Characteristics
* At least 1 week since prior tamoxifen
* No concurrent anticancer hormonal therapy
* See Disease Characteristics
* No concurrent anticancer radiotherapy
* See Disease Characteristics
* Prior recent resection of recurrent or progressive tumor allowed if patient has recovered
* Recovered from all prior therapy
* At least 2 weeks since prior EIAEDs (patients in Group A only)
* At least 4 weeks since prior cytotoxic therapy
* At least 4 weeks since prior investigational agents
* At least 1 week since prior isotretinoin
* At least 1 week since other prior non-cytotoxic therapy (except radiosensitizers)
* No concurrent valproic acid
* No concurrent hydrochlorothiazide
* No concurrent medication that causes QTc prolongation
* No other concurrent anticancer therapy
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-01; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Fine, MD, Principal Investigator — North American Brain Tumor Consortium
Locations (8):
- United States (8):
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - National Cancer Institute Neuro-Oncology Branch, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iwamoto FM, Lamborn KR, Kuhn JG, Wen PY, Yung WK, Gilbert MR, Chang SM, Lieberman FS, Prados MD, Fine HA. A phase I/II trial of the histone deacetylase inhibitor romidepsin for adults with recurrent malignant glioma: North American Brain Tumor Consortium Study 03-03. Neuro Oncol. 2011 May;13(5):509-16. doi: 10.1093/neuonc/nor017. Epub 2011 Mar 3. PMID 21377994

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Escalation - Romidepsin: Patients receive FR901228 (romidepsin) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Dose escalation two dose levels:
  Romidepsin (depsipeptide): 13.3mg/m2 and 17.7mg/m2
  Pharmacokinetics
  depsipeptide: Given IV
- Phase 2 Dose From Phase 1 - Romidepsin: Patients receive FR901228 (romidepsin) as in phase I at dose level 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Romidepsin (depsipeptide): 13.3mg/m2
  depsipeptide: Given IV
Period: Overall Study
Arm/Group | Phase 1 Dose Escalation - Romidepsin | Phase 2 Dose From Phase 1 - Romidepsin
Started | 8 | 42
Completed | 8 | 40
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: two patients were removed from the analysis due to one withdrawing consent and one was deemed ineligible.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Escalation - Romidepsin | Phase 2 Dose From Phase 1 - Romidepsin | Total
Number analyzed (Participants) | 8 | 40 | 48
Age, Continuous [Median (Full Range); unit: years] | 52 [44 to 57] | 55 [37 to 79] | 54 [37 to 79]
Gender [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 5 | 30 | 35
Karnofsky Performance Status Scale (KPS) [Number; unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale
    90-100 | 4 | 19 | 23
    60-80 | 4 | 21 | 25
Histology [Number; unit: participants]
  Anaplastic glioma | 2 | 5 | 7
  Gliobastoma | 6 | 35 | 41
Prior Radiotherapy [Number; unit: participants] | 8 | 40 | 48
Prior chemotherapy regimens [Median (Full Range); unit: number of chemotherapy regimens] | 1 [1 to 2] | 1 [1 to 3] | 1 [1 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities Due to Romidepsin Graded According to the NCI Common Toxicity Criteria (CTCAE Version 3.0) (Phase I)
Description: dose limiting toxicity defined as: ANC </=1000 or Platelets <100K; SGOT >/= 3X ULN and T. Bili >/= 1.5 ULN
  grade 3 Nausea, vomiting, fatigue and asymptomatic hypocalcemia (treatment may continue after discuss with PI)
Time Frame: First 4 weeks of treatment
Measure: Number; unit: participants
Arm/Group | Phase 1 Dose Escalation - Romidepsin
Number analyzed (Participants) | 8
participants | 0

2. Primary Outcome: 6 Months Progression-free Survival (Phase II)
Description: evaluated patients with glioblastoma (GBM (35 patients)
Time Frame: At 6 months
Population: evaluation of patients with GBM histology
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2 Dose From Phase 1 - Romidepsin
Number analyzed (Participants) | 35
percentage of participants | 3

3. Secondary Outcome: Response Rate Associated With Depsipeptide Therapy (Phase II)
Description: RECIST Complete Response (CR): Complete disappearance of all measurable and evaluable disease. No new lesions. No evidence of non-evaluable disease. Patients must be on no steroids.
  Partial Response (PR): Greater than or equal to 50% decrease under baseline in the sum of products of perpendicular diameters of all measurable lesions. No progression of evaluable disease. No new lesions.
  Stable/No Response: Does not qualify for CR, PR, or progression. The designation of Stable/No Response requires a minimum of 8 weeks duration.
  Progression: 25% increase in the sum of products of all measurable lesions over smallest sum observed (over baseline if no decrease) OR clear worsening of any evaluable disease, OR appearance of any new lesion/site, OR clear clinical worsening or failure to return for evaluation due to death or deteriorating condition
Time Frame: Up to 2 years
Population: GBM patients - no responses
Measure: Number; unit: participants
Arm/Group | Phase 2 Dose From Phase 1 - Romidepsin
Number analyzed (Participants) | 35
participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Description: in the phase 1 portion of the study the DLT were reviewed in the first 4 weeks only
Arm/Group | Phase 1 Dose Escalation - Romidepsin | Phase 2 Dose From Phase 1 - Romidepsin
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/40
Other Adverse Events (participants affected / at risk) | 8/8 | 40/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Escalation - Romidepsin (N=8) | Phase 2 Dose From Phase 1 - Romidepsin (N=40)
anemia (Blood and lymphatic system disorders) | 3 (3) | 8 (8)
Leucopenia (Blood and lymphatic system disorders) | 3 (3) | 8 (8)
neutropenia (Blood and lymphatic system disorders) | 3 (3) | 7 (7)
lymphopenia (Investigations) | 1 (1) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6) | 15 (15)
Alkaline phosphatase elevation (Investigations) | 1 (1) | 1 (1)
elevated ALT and/or AST (Investigations) | 2 (2) | 9 (9)
anorexia (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
hypogycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
fatigue (General disorders) | 4 (4) | 17 (17)
muscle weakness (lower extremity) (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
headache (Nervous system disorders) | 4 (4) | 1 (1)
hot flashes (Vascular disorders) | 1 (1) | 0 (0)
gait disturbance (General disorders) | 1 (1) | 0 (0) — gait or walking difficulties
nausea (Gastrointestinal disorders) | 5 (5) | 13 (13)
rigors or chills (General disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
constipation (Gastrointestinal disorders) | 0 (0) | 7 (7)
diarrhea (Gastrointestinal disorders) | 0 (0) | 4 (4)
heartburn (Gastrointestinal disorders) | 0 (0) | 2 (2)
edema-limb (General disorders) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Dose escalation was terminated after 2 dose levels because PK parameters of romidepsin in pts receiving EIAEDs were similar to those reported in Adults not receiving CYP34A inducing drugs, we wanted to avoid the expected dose limiting toxicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less